CLINICAL TRIAL: NCT01674322
Title: An Open-Label Phase 1 Study to Determine the Pharmacokinetics, Metabolism, and Routes of Excretion of (14C) Radiolabeled PCI-32765 in Healthy Male Subjects
Brief Title: A Study to Determine the Absorption, Metabolism, and Routes of Excretion of (14C) Radiolabeled Ibrutinib in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100885; PCI-32765CLL1004 (Other: Janssen Research & Development, LLC); 2012-002087-27 (EudraCT Number)
Record Dates: First submitted 2012-08-09; First posted 2012-08-28 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Participants
Keywords: Healthy participants; Ibrutinib; PCI-32765; B-cell malignancies; CYP3A4
MeSH Terms: interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ibrutinib (Experimental): All participants will receive a single oral solution dose of 50 mg to 140 mg -ibrutinib containing 1480 kBq (40 µCi) of 14C-labeled ibrutinib, with a total radiation burden of approximately 0.916 mSv.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Type=exact number, unit=mg, number=50-140, form=solution, route=oral. Participants will receive a single oral solution dose of 50 mg to 140 mg -ibrutinib containing 1480 kBq (40 µCi) of 14C-labeled ibrutinib, with a total radiation burden of approximately 0.916 mSv.
  Other Names: PCI-32765

SUMMARY:
The purpose of this study is to investigate the absorption, the metabolic pathways and the excretion of ibrutinib in healthy male adult participants after administration of a single oral dose of 50 mg to 140 mg (5 mg/mL solution) of unlabeled ibrutinib admixed with 14C ibrutinib.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-center, single-dose study in healthy male participants. Six men will be enrolled to allow a minimum of 4 participants to complete the study. All participants will receive a single oral solution dose of 50 to 140 mg ibrutinib containing 1480 kBq (40 µCi) of 14C labeled ibrutinib, constituting a total radiation burden of approximately 0.916 mSv (ICRP risk category IIa). The duration of the study is approximately 73 days including screening period of 28 days, treatment period of 15 days, and follow-up period of 30 days. Safety will include adverse events, laboratory safety, 12 lead electrocardiogram, physical examination, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Participant must sign an informed consent document indicating they understand the purpose of and procedures required for the study, including DNA analysis, and are willing to participate in the study
* Must agree to use an adequate contraception method as deemed appropriate by the investigator (eg, vasectomy, double-barrier, partner using effective contraception) during the study and for 3 months after receiving the study drug
* Must agree to not donate sperm during the study and for 3 months after receiving the study drug
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic
* Non-smoker (not smoked for 6 months prior to screening)

Exclusion Criteria:

* History of or current clinically significant medical illness including cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders, lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease
* Clinically significant abnormal values for hematology, coagulation and platelet function, clinical chemistry or urinalysis at screening as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs or 12 lead electrocardiogram (ECG) at screening as deemed appropriate by the investigator
* History of clinically significant allergies, especially known hypersensitivity or intolerance to β-lactam antibiotics or sulfonamides
* Known allergy to heparin or history of heparin induced thrombocytopenia

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of ibrutinib | Day 1 (Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 hours), Day 2 (24 hours), Day 3 (48 hours), Day 4 (72 hours)
  Pharmacokinetic parameter Cmax of ibrutinib will be determined.
Time to reach the maximum concentration (tmax) of ibrutinib | Predose, Day 1 (0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 hours), Day 2 (24 hours), Day 3 (48 hours), Day 4 (72 hours)
  Pharmacokinetic parameter tmax of ibrutinib will be determined.
Area under the concentration-time curve (AUC) of ibrutinib | Predose, Day 1 (0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 hours), Day 2 (24 hours), Day 3 (48 hours), Day 4 (72 hours)
  Pharmacokinetic parameter AUC of ibrutinib will be determined.
Amount excreted into the urine (Ae) of ibrutinib | Day -1, Day 1 over intervals 0-2, 2-4, 4-8, 8-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168 hours, Days 9-15
  Pharmacokinetic parameter Ae of ibrutinib will be determined by multiplying the urinary volume with the urinary concentration.

SECONDARY OUTCOMES:
Number of patients with adverse events | Up to 73 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium

REFERENCES:
- [Derived] Scheers E, Leclercq L, de Jong J, Bode N, Bockx M, Laenen A, Cuyckens F, Skee D, Murphy J, Sukbuntherng J, Mannens G. Absorption, metabolism, and excretion of oral (1)(4)C radiolabeled ibrutinib: an open-label, phase I, single-dose study in healthy men. Drug Metab Dispos. 2015 Feb;43(2):289-97. doi: 10.1124/dmd.114.060061. Epub 2014 Dec 8. PMID 25488930